CLINICAL TRIAL: NCT01791699
Title: Pharmacologic Suppression of Central Sympathetic Activity for Prevention of Atrial Fibrillation Recurrence After Pulmonary Vein Isolation (MOXAF)
Brief Title: Moxonidine for Prevention of Post-ablation AFib Recurrences
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Spyridon Deftereos (Other)
Responsible Party: Sponsor-Investigator, Spyridon Deftereos, Director; Catheterization Laboratory and Cardiac Electrophysiology Laboratory, G.Gennimatas General Hospital
Organization: G.Gennimatas General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOX.AFABL.9.5.2012
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; paroxysmal; persistent; ablation; pulmonary vein isolation; recurrence
MeSH Terms: conditions — Atrial Fibrillation; Recurrence | interventions — moxonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator): The patients of the control group will undergo standard ablation procedure (pulmonary vein isolation) and will receive placebo, starting one week before scheduled ablation.
  Optimal antihypertensive treatment will be prescribed, with adequate follow-up to ensure good control of hypertension (goal <= 140/90).
  Interventions: Drug: Placebo
- Moxonidine group (Active Comparator): Patients of the active treatment group will receive moxonidine in a starting dose of 0.2 mg daily. The first dose will be administered 1 week before scheduled ablation. 3 weeks after the first dose the daily dose will be increased to 0.4 mg, if the lower dose is well tolerated.
  Optimal antihypertensive treatment, in addition to moxonidine, will be prescribed, if needed, with adequate follow-up to ensure good control of hypertension (goal <= 140/90).
  Interventions: Drug: Moxonidine

INTERVENTIONS:
Drug: Moxonidine
  Arms: Moxonidine group
Drug: Placebo
  Arms: Control group

SUMMARY:
Hypothesis: Modulation of central nervous sympathetic activation by administration of moxonidine, a centrally acting medication which decreases the sympathetic nervous system activity, can lead to a decrease in atrial fibrillation recurrence after ablation treatment with pulmonary vein isolation.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients with paroxysmal atrial fibrillation.
* At least two documented episodes within the last 12 months (either self-terminating within 7 days or cardioverted, medically or electrically, in less than 48 hours).
* At least one episode should have been documented under treatment with a class Ic or III antiarrhythmic drug.

Exclusion Criteria:

1. age <25 or >80 years
2. presence of atrial thrombus
3. left atrial volume index >55 ml/m2
4. hypersensitivity to moxonidine
5. sick sinus syndrome or sino-atrial block
6. 2nd or 3rd degree atrioventricular block
7. bradycardia (below 50 beats/minute at rest)
8. estimated glomerular filtration rate <40 ml/min/1.73 m2
9. history of angioneurotic oedema
10. heart failure symptoms OR impaired left ventricular function (EF <40%), even if asymptomatic
11. stable or unstable angina pectoris
12. intermittent claudication or known peripheral artery disease
13. Parkinson's disease
14. epileptic disorders
15. glaucoma
16. history of depression
17. pregnancy or lactation
18. inability or unwillingness to adhere to standard treatment or to provide consent.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
AFib recurrence | 12 months+
  Any of the following, occuring after a 3-month blanking period, will be considered an AF recurrence:
  * symptomatic recurrence (AF/MRAT of any duration in ECGs performed in patients reporting symptoms of arrhythmia); the patients will be encouraged to visit the research site or any affiliated center to have an ECG performed at any time (24/7) they may feel symptoms of arrhythmia during the study follow-up
  * AF/MRAT of at least 30 seconds in duration in 48-hour Holter recordings performed monthly
  * AF/MRAT of any duration recorded in electrocardiograms performed during patient visits at the arrhythmia clinic, even if the patient is asymptomatic
  (AF=atrial fibrillation, MRAT=macro-reentrant atrial tachycardia)

SECONDARY OUTCOMES:
Depressive symptoms | 6 months
  The 17-item Hamilton Depression Rating Scale will be administered at baseline, and at the 3- and 6-month visits.
Early AFib recurrence | 2 months
  Any of the following, occuring within 2 months post-ablation, will be considered an early AF recurrence:
  * symptomatic recurrence (AF/MRAT of any duration in ECGs performed in patients reporting symptoms of arrhythmia); the patients will be encouraged to visit the research site or any affiliated center to have an ECG performed at any time (24/7) they may feel symptoms of arrhythmia during the study follow-up
  * AF/MRAT of at least 30 seconds in duration in 48-hour Holter recordings performed monthly
  * AF/MRAT of any duration recorded in electrocardiograms performed during patient visits at the arrhythmia clinic, even if the patient is asymptomatic

OTHER OUTCOMES:
Adverse effects | 6 months
  Moxonidine-related adverse effects will be monitored and recorded, focusing on xerostomia, headaches, sleep disorders, hypotension, orthostatic hypotension

CONTACTS AND LOCATIONS:
Locations (3):
- Greece (3):
  - Evangelismos General Hospital, Athens
  - Athens General Hospital "G. Gennimatas", Athens
  - Red Cross Hospital, Athens

REFERENCES:
- [Derived] Giannopoulos G, Vrachatis D, Kossyvakis C, Angelidis C, Koutivas A, Tsitsinakis G, Zacharoulis A, Kolokathis F, Palaiologos D, Vavuranakis M, Deftereos S. Effect of Postablation Statin Treatment on Arrhythmia Recurrence in Patients With Paroxysmal Atrial Fibrillation. J Cardiovasc Pharmacol. 2018 Dec;72(6):285-290. doi: 10.1097/FJC.0000000000000624. PMID 30520854
- [Derived] Giannopoulos G, Kossyvakis C, Angelidis C, Efremidis M, Panagopoulou V, Letsas K, Bouras G, Vassilikos VP, Goudevenos J, Tousoulis D, Lekakis J, Deftereos S. Amino-terminal B-natriuretic peptide levels and postablation recurrence in hypertensive patients with paroxysmal atrial fibrillation. Heart Rhythm. 2015 Jul;12(7):1470-5. doi: 10.1016/j.hrthm.2015.04.002. Epub 2015 Apr 3. PMID 25847478
- [Derived] Giannopoulos G, Kossyvakis C, Efremidis M, Katsivas A, Panagopoulou V, Doudoumis K, Raisakis K, Letsas K, Rentoukas I, Pyrgakis V, Manolis AS, Tousoulis D, Stefanadis C, Deftereos S. Central sympathetic inhibition to reduce postablation atrial fibrillation recurrences in hypertensive patients: a randomized, controlled study. Circulation. 2014 Oct 14;130(16):1346-52. doi: 10.1161/CIRCULATIONAHA.114.010999. Epub 2014 Aug 21. PMID 25147079